CLINICAL TRIAL: NCT06736821
Title: Clinical, Radiographic and Histomorphometric Assessment of the Effect of Melatonin Gel Mixed With Xenograft in Augmentation of the Maxillary Sinus: A Randomized Controlled Clinical Trial
Brief Title: Maxillary Sinus Augmentation by Xenograft Mixed With Melatonin
Acronym: melatonin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: rehab soliman (Other)
Responsible Party: Sponsor-Investigator, rehab soliman, lecturer of oral and maxillofacial department, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 710/2023
Record Dates: First submitted 2024-12-08; First posted 2024-12-17 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Bone Healing
Keywords: sinus lifting; maxillary sinus augmentation; melatonin gel
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: This study was included16 severely atrophied maxillary sinus, with alveolar bone height less than 4mm, that need sinus augmentation and delayed implant placement. all patients was enrolled randomly and distributed into 2 groups (via : http://www.randomizer.org) :
  Group A: sinus membrane elevation was done using lateral window technique and filled with the mixture of melatonin and xenograft.
  Group B: sinuses membrane was elevated and filled with with xenograft. After 6 months, bone biopsies was collected from the augmented sinuses immediately before implant instalment in the same visit.
  Initial CBCT was taken preoperatively and immediate postoperatively. Final CBCT was taken 6 months before implant placement to measure Bone density and bone height and width.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group a: xenograft mixed with melatonin (Experimental): in this group, the patients underwent open sinus lifting surgery and augmentation of the sinuses by xenograft mixed with melatonin gel to enhance the bone healing
  Interventions: Dietary Supplement: Open sinus augmentation with melatonin gel mixed with xenograft
- group b: xenograft (Active Comparator): in this group, the patients underwent open sinus lifting surgery and augmentation of the sinuses by xenograft without any additives
  Interventions: Procedure: Open sinus augmentation with xenograft

INTERVENTIONS:
Dietary Supplement: Open sinus augmentation with melatonin gel mixed with xenograft — All Patients in this group underwent open sinus procedures to lift the sinus membrane followed by application of the melatonin gel which was mixed with xenograft as an augmentation material.
  Preclinical studies proved the direct action of melatonin in enhancing the differentiation and proliferation of bone-forming osteoblasts. In addition to increasing bone mass, melatonin also facilitates new bone growth and osteointegration, making melatonin a particularly attractive molecule for use in bone implants when used alone or in combination with other growth factors
  Other Names: Primary intervention
  Arms: group a: xenograft mixed with melatonin
Procedure: Open sinus augmentation with xenograft — All Patients in this group underwent open sinus procedures to lift the sinus membrane followed by application of the xenograft as an augmentation material xenograft is used instead of autogenous bone graft to avoid the morbidity of the donor side
  Other Names: Secondary Intervention
  Arms: group b: xenograft

SUMMARY:
The possibility of enhancing the bone substitute in the maxillary sinus by mixing it with the melatonin to allow proper implant placement in early stage .

The aim of the study was to evaluate clinically, radiographically and histologically the effect of melatonin in enhancement of bone healing after augmentation of the maxillary sinus.

DETAILED DESCRIPTION:
This study was include 16 severely atrophied maxillary sinus, with alveolar bone height less than 4mm, that need sinus augmentation and delayed implant placement, they were be equally and randomly distributed into 2 groups (via : http://www.randomizer.org) :

Group A: sinuses was received sinus membrane elevation using lateral window technique and filling the sinus with the mixture of melatonin and xenograft.

Group B: sinuses was received sinus membrane elevation using lateral window technique and filling the sinus with xenograft.

After 6 months, bone biopsies was collected from the augmented sinuses immediately before implant instalment in the same visit.

Initial cone beam computerized tomography was taken preoperatively and immediate postoperatively.

Final cone beam computerized tomography was taken 6 months before implant placement to measure Bone density and bone height and width.

After 3 months of implant placement, the installed implants was assessed clinically to exclude any infection or dehiscence and radio graphically to assess the bone loss or any radiolucent lesion around the implants and then prepared for loading.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female patients above the age of 25.
2. Patients with one or more teeth requiring implant supported dental restoration in atrophic maxilla (unilateral or bilateral).
3. Alveolar bone height less than 4 mm at the defective site.
4. Good oral hygiene.

Exclusion Criteria:

1. Medically compromised patients with conditions contraindicating surgery (eg. uncontrolled diabetics, bisphosphonate intake, radio or chemotherapy).
2. Patients with active infection at or related to the site of surgery (eg. acute sinusitis).
3. Heavy smokers.
4. Patients not indicated for an implant supported restoration at the time of enrollment (eg. active/untreated periodontal disease).

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Alveolar Bone Height | 8 months
  Alveolar Bone height was measured using cone beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Histological Analysis of Newly Formed Bone | 8 months
  The quality of the newly formed bone was evaluated using two histological stains: Hematoxylin and Eosin, and Masson's Trichrome.

CONTACTS AND LOCATIONS:
Overall Officials: rehab soliman, Principal Investigator — Misr International University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No